CLINICAL TRIAL: NCT02435316
Title: A Randomized, Controlled Cross Over Trial of Two Educational Methods and Their Additive Effects in the Recognition of Abnormal Peripheral Blood Smears
Brief Title: Comparison of Educational Methods for Teaching Peripheral Blood Smears
Acronym: PBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Reading Hospital and Medical Center (Other)
Responsible Party: Principal Investigator, Anthony A. Donato, Associate Program Director, Inpatient Medicine, The Reading Hospital and Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TRHMC 016-12
Record Dates: First submitted 2015-04-30; First posted 2015-05-06 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Hematologic Diseases
Keywords: Education
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 will receive 1 hour of compare-contrast basic science teaching of cell recognition to enhance recognition of those photographs, followed by 1 hour Case vignette-based teaching of cell recognition 2 weeks later
  Interventions: Other: Case vignette-based teaching of cell recognition; Other: Compare-contrast basic science teaching of cell recognition
- Group 2 (Active Comparator): Group 2 will receive 1 hour of Case vignette-based teaching of cell recognition followed by compare-contrast basic science teaching of cell recognition 2 weeks later
  Interventions: Other: Case vignette-based teaching of cell recognition; Other: Compare-contrast basic science teaching of cell recognition

INTERVENTIONS:
Other: Case vignette-based teaching of cell recognition — Intervention group members will be taught peripheral blood smears by using power point slides and utilizing additive microskills using the compare/ contrast technique to recognize various cell types. Memory will be reinforced by using cases to help recognize the clinical importance of learning about individual cell types.
Other: Compare-contrast basic science teaching of cell recognition — The control group will be given a traditional 60-minute lecture using board review questions with accompanying pictures of peripheral blood smears, without explaining individual cell type.

SUMMARY:
This is a prospective, randomized controlled, crossover trial comparing the effectiveness one two curricular designs to teaching peripheral blood smears to residents.

DETAILED DESCRIPTION:
General Approach:

This study will employ a randomized, controlled design and will use as its outcomes two separate post-tests, one after the first teaching session and one 4 weeks after the second intervention.

Design The investigators are attempting to find whether the combination of basic science education using an 1-hour additive microskills- building method along with compare/ contrast model versus a 1-hour traditional case-based format would improve performance on a visual recognition test of hematology questions. A final test at 4 weeks after the cross-over between the two groups will also help investigators analyze whether the order of exposure to the teaching method would have an impact on the final performance.

Sampling, including sample size and statistical power:

Sample size will be between 40-50 resident physicians meeting inclusion criteria for the study. There is not enough data in the literature to effectively determine power, so we will use a convenience sample of the largest feasible group (around 40).

Collection of data:

Data will be collected on an excel spreadsheet and will be permanently de-identified on that spreadsheet; it will be kept on a password-protected site.

Information management and analysis software:

Data will be entered into a password protected excel spreadsheet and each study participant will be assigned a unique identifier code which will be used to link the data. Statistical analysis will be performed using SPSS version 20.

Data entry, editing and management, including handling of data collection forms, different versions of data, and data storage and disposition:

Paper surveys and tests will be collected, recorded and locked; they will be destroyed 2 years after termination of the study. A paired t-test will be used to compare the two samples means for significance.

Quality Control / Assurance:

Pretest and post-tests will be checked against a gold standard, a hospital board-certified hematopathologist, to check the quality of the slides.

Bias in data collection, measurement and analysis:

Given the small numbers of participants expected, a Type 1 error (failure to detect a difference in groups when one exists) is possible, as the study will possibly be underpowered.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine and Family Medicine residents and faculty at The Reading Hospital and Medical Center having completed medical school

Exclusion Criteria:

* Practicing/ board certified hematologists

Ages: 26 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2013-02-12 (Actual)

PRIMARY OUTCOMES:
Improvement in post test scores at 2 and 4 weeks after education | 4 weeks
  Primary outcome was an improvement in test score from pre-test to 2 and 4-week post-test. All participants took a 15-question pretest in addition to a posttest at 2 and 4 weeks. Each test consisted of pictures of various cell types from the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Donato, MD, Study Director — The Reading Hospital and Medical Center
Locations (1):
- Reading Health System, West Reading, Pennsylvania, United States